CLINICAL TRIAL: NCT07148050
Title: Immunotherapy for Solid Tumor Malignancies in Pediatrics Using Interleukin-15 and -21 Armored Glypican-3-specific Chimeric Antigen Receptor T Cells
Acronym: IMPACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director - Seattle Children's Therapeutic, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor (Excluding CNS); Liver Cell Carcinoma; Malignant Rhabdoid Tumor; Yolk Sac Tumor; Liposarcoma; Rhabdomyosarcoma; Embryonal Sarcoma of Liver; Wilms Tumor; Hepatocellular Carcinoma; Hepatoblastoma
Keywords: CAR T cell; Pediatric; Young Adult; Non-CNS Tumor; Liver Cancer; Solid Tumor; GPC3; Glypican
MeSH Terms: conditions — Carcinoma, Hepatocellular; Rhabdoid Tumor; Endodermal Sinus Tumor; Liposarcoma; Rhabdomyosarcoma; Wilms Tumor; Hepatoblastoma; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SC-CAR.GPC3xIL15.21 T cells (Experimental): Autologous SC-CAR.GPC3xIL15.21 T cell product will be infused as a single infusion.
  Interventions: Biological: SC-CAR.GPC3xIL15.21 CAR T cells

INTERVENTIONS:
Biological: SC-CAR.GPC3xIL15.21 CAR T cells — Autologous SC-CAR.GPC3xIL15.21 T cell products infusion

SUMMARY:
This Phase 1, open-label, non-randomized study will enroll pediatric and young adult subjects with relapsed or refractory non-central nervous system (CNS) malignant solid tumors expressing glypican-3 (GPC3) to examine the safety, feasibility, and efficacy of administering T cell products derived from peripheral blood mononuclear cells (PBMC) that have been genetically modified to co-express a GPC3-specific chimeric antigen receptor (CAR), interleukin (IL)-15 and IL-21 as well as the inducible caspase 9 (iC9) suicide gene (SC-CAR.GPC3xIL15.21 T cells).

A child or young adult meeting all eligibility criteria and meeting none of the exclusion criteria will have a blood sample collected, which will be used to bioengineer the CAR T cells targeting their tumor.

DETAILED DESCRIPTION:
Study Overview

This study is testing a different treatment which uses the body's own immune system to recognize and kill the cancer cells, called chimeric antigen receptor (CAR) T cells. Some solid tumors express a specific type of molecule called glypican-3 or GPC3. We are able to insert a new gene (a piece of DNA that contains a set of instructions for the body) into T cells which are a type of immune system cell. This is how we make CAR T cells: We will insert a gene that will program the CAR T cell to recognize GPC3 to make GPC3-CAR T cells. To make GPC3-CAR T cells more effective against tumor cells, we also added two genes called IL15 and IL21 which help CAR T cells grow better and stay in the blood longer. We think that this will kill tumors better. When we did this in the laboratory, we found that this mixture of GPC3-CAR, IL15, and IL21 in T cells killed tumor cells better when compared with GPC3-CAR T cells that did not have IL15 and IL21. This research study will use these cells (named GPC3xIL15.21) to treat patients with solid tumors that express GPC3 on their surface. The GPC3xIL15.21 CAR T cells are an investigational product and have not been approved by the Food and Drug Administration.

We also wanted to make sure that we could stop the GPC3xIL15.21 CAR T cells from growing in the blood if there are any bad or severe side effects. To do so, we inserted a gene called iCasp9 into the GPC3xIL15.21 CAR T cells. This allows us to eliminate the GPC3xIL15.21 CAR T cells in the blood when we give a medicine called AP1903 (also known as rimiducid). Rimiducid is an experimental medicine that has been tested in humans, with no known bad side effects. We only intend to use this medicine to get rid of the GPC3xIL15.21 CAR T cells if you develop dangerous side effects. Approximately 21 people will participate in this study.

Treatment plan

We would first confirm that the participant tumor expresses GPC3. Upon confirmation, a maximum of approximately 6 tablespoons (or 90 mL) of blood will be drawn and sent to Seattle Children's Therapeutics (SCTx) to make the CAR T cells.

After the CAR T cells are made and treatment eligibility has been verified, participants will come to Seattle Children's Hospital for treatment and close monitoring for about one month. Participants will be given lymphodepleting chemotherapy for 3 days, using cyclophosphamide and fludarabine to make room for the CAR T cells, followed by CAR T cell infusion IV.

This is a dose escalation study, which means that the investigators do not know the highest safe dose of CAR T cells. The dose each patient gets depends on how many participants get the agent before that patient and how they react. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the treatments will be given at Seattle Children's Hospital.

After treatment, participants will be monitored closely for a month to monitor for side effects and response to treatment. After this month, participants would continue to be followed for 15 years after they receive your CAR T cells, with visits becoming less frequent the longer it has been since CAR T cell infusion.

ELIGIBILITY:
1. Procurement Eligibility

   Inclusion Criteria:
   * Diagnosis of a solid tumor expressing GPC3
   * Lansky or Karnofsky score of >=60%
   * Life expectancy of >16 weeks
   * Informed consent explained to, understood by and signed by patient/guardian.

   For patients with hepatocellular carcinoma only:
   * Barcelona Liver Cancer Stage A, B or C
   * Child-Pugh Turcotte Score <7

   Exclusion Criteria:
   * History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies.

     * History of organ transplantation
     * Known HIV positivity
     * Active bacterial, fungal, or viral infection (except Hepatitis B or Hepatitis C virus infections)
2. Treatment eligibility

Inclusion Criteria:

* Lansky or Karnofsky score of >=60%
* Life expectancy of >16 weeks
* Informed consent explained to, understood by and signed by patient/guardian.
* Adequate organ function
* Adequate laboratory values
* Refractory or relapsed disease after treatment with up- front therapy and at least one salvage treatment cycle
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 12 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/guardian.

For patients with hepatocellular carcinoma only:

* Barcelona Liver Cancer Stage A, B or C
* Child-Pugh Turcotte Score <7

Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies.

  * History of organ transplantation
  * Known HIV positivity
* Active autoimmune or inflammatory disorder
* Live vaccines within 30 days prior to enrollment

  • Active bacterial, fungal, or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Pregnancy or lactation
* Uncontrolled infection
* Systemic steroid treatment (≥ 0.5 mg prednisone equivalent/kg/day, dose adjustment or discontinuation of medication must occur at least 24hrs prior to CAR T cell infusion)
* Congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2029-04-22 (Estimated); Study Completion 2044-04-22 (Estimated)

PRIMARY OUTCOMES:
The number of successfully manufactured SC-CAR.GPC3xIL15.21 T cell products will be assessed | 28 days
  The number of successfully manufactured products will be measured
Establish the safety, defined by adverse events of SC-CAR.GPC3xIL15.21 T cells. | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized

SECONDARY OUTCOMES:
Estimate the maximum tolerated dose (MTD) or biologically effective dose and dose limiting toxicities (DLT), and describe the full toxicity profile of SC-CAR.GPC3xIL15.21 T cells. | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To estimate anti-tumor responses by measuring changes in tumor burden using disease-specific evaluations following SC-CAR.GPC3xIL15.21 T cells. | 42 days
  Standard imaging and blood pathology will be used to determine disease response

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Director — Seattle Children's Hospital; Corinne Summers, MD, Study Director — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No